CLINICAL TRIAL: NCT06141668
Title: Optimal Stimulation Parameters for Spike-ripple Disruption in Patients Undergoing Invasive Monitoring
Brief Title: Optimal Stimulation Parameters to Disrupt Epileptiform Activity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Boston University (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Catherine Chu, MD, Associate Professor Neurology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 2020P002398; R01NS119483 (NIH)
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Refractory Epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Neurostimulation — Electrical stimulation

SUMMARY:
Open-loop electrical stimulation has been found to reduce spike activity and seizures, but determining the optimal parameters to achieve these effects requires a brute force trial-and-error approach that relies on subjective physician discretion. We will compare the performance of stimulation parameters identified in rodent models to the recommended parameters for neuromodulation used in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

- Undergoing intracranial EEG investigation at Massachusetts General Hospital during presurgical epilepsy evaluation

Exclusion Criteria:

- Baseline spike ripple rate < 0.5/min.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Spike ripple rate | 1-3 hours

SECONDARY OUTCOMES:
Spike rate | 1-3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Chu, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No